CLINICAL TRIAL: NCT03314415
Title: Pilot Study on Weight Loss With Robotic Assistance
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study will not be implemented and did not enroll participants.
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Susan Roberts, Director and Senior Scientist, Tufts University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12561
Record Dates: First submitted 2017-07-17; First posted 2017-10-19 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Overweight and Obesity; Weight Loss
Keywords: overweight; obesity; weight loss; robot
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Robotic-assisted weight loss
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early robotic intervention (Experimental): Participants randomized to the early robotic intervention will attend robotic assistance sessions for a two-week period earlier in the study (during the first half of the study, approximately). Each participant will attend ten 15-minute robotic assistance sessions to interact with a robot (Aldebaraan Nao H25).
  Interventions: Device: Aldebaraan Nao H25
- Late robotic intervention (Experimental): Participants randomized to the late robotic intervention will attend robotic assistance sessions for a two-week period later in the study (during the latter half of the study, approximately). Each participant will attend ten 15-minute robotic assistance sessions to interact with a robot (Aldebaraan Nao H25).
  Interventions: Device: Aldebaraan Nao H25

INTERVENTIONS:
Device: Aldebaraan Nao H25 — The Aldebaraan Nao H25 is a humanoid robot with the capability to interact with people through small movements, gestures, and speech. It does not physically touch the participant at any time.

SUMMARY:
The purpose of this study is to determine whether robotic assistance can help facilitate adherence, engagement, and weight loss in participants enrolled in a behavioral weight loss program. All participants will be enrolled in the same Web-based weight loss program and take part in "robotic assistance sessions" either early or late in the five-week study. These robotic assistance sessions involve speaking one on one with a robot about diet-related progress.

DETAILED DESCRIPTION:
At the start of the five-week study, all participants will be enrolled in a Web-based behavioral weight loss program. The weight loss program places particular emphasis on hunger reduction and craving control for both weight loss and prevention of weight regain. The program will consist of six videoconference sessions delivered by a qualified coach. Menus and other program materials will be available to the participants throughout the study period.

Participants also will be assigned to attend one-on-one "robotic assistance sessions" either early or late in the five-week study. During each robotic assistance session, the participant will speak with the robot about his/her progress with the weight loss program. The robot is programmed to respond to specific issues raised by the participant, but a human operator with thorough knowledge of the weight loss program will be available in case the conversation goes "off script." This human operator can initiate robot behaviors and prompt verbal responses through a text-to-speech interface.

Data from this study will be used to refine the robot for future use and determine whether robotic help can improve a participant's experience in a previously tested weight loss program.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are overweight or obese (body mass index of 25-40 kg/m2)
* Want to lose weight and enroll in the study, and are willing to sign the informed consent form
* Able to meet the study requirements for food habits and able to attend online videoconference sessions
* Willing and able to attend in-person robotic assistance sessions, and are not planning to be out of town for more than five days during the study

Exclusion Criteria:

* Self-reported serious food allergies/intolerances, dietary patterns, or active health conditions (e.g., irritable bowel syndrome, Crohn's disease, celiac disease) that would prevent consumption of recommended foods.
* Concurrent participation in another weight loss program or >2 hours/day of exercise on average.
* Actively dieting or self-reported weight loss of >10 lb in the past 3 months
* Vulnerable populations, including women who are pregnant and adults who are unable to consent
* Women who are lactating or planning to become pregnant within two months of the start date, per self-report
* Diagnosis of a serious mental health condition
* Non-English speaking individuals
* Medical complications or chronic illness that would prevent full participation (e.g., active cancer)
* Surgical procedures that influence hunger or satiety (e.g., gastric bypass, bowel rerouting, stomach sleeve)
* Primary training as a Clinical Nutritionist or practicing Registered Dietitian
* Diagnosed eating disorder

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-11 (Estimated); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Weight change | 5 weeks
  Primary outcome is weight change during the with-robot and without-robot periods adjusted for week of weight loss.

SECONDARY OUTCOMES:
Change in self-reported eating behavior | Baseline, once during with-robot phase, Week 5
  Participants will complete the Three-Factor Eating Questionnaire, consisting of 18 items, which will be used to assess eating behavior on a 4-point response scale (4=definitely true;3=mostly true;2=mostly false;1=definitely false). Responses to each of the 18 items are given a score between 1 and 4 and item scores are summed into scale scores for cognitive restraint, uncontrolled eating, and emotional eating. Total scores will be reported and higher scores in the respective scales are indicative of greater cognitive restraint, uncontrolled, or emotional eating. Questionnaires are self-administered.
Change in self-reported food cravings | Baseline, once during with-robot phase, Week 5
  Participants will complete the Food Cravings Questionnaire - Trait, which will be used to assess food cravings on a 6-point response scale (1=Never or NA;2=Rarely; 3=Sometimes;4=Often;5=Usually;6=Always). Responses to each of the 39 items are given a score between 1 and 6 and item scores are summed into scale scores with higher scores being indicative of greater eating pathology, body mass index (BMI), low dieting success and increases in state food craving during cognitive tasks. Total scores will be reported. Questionnaires are self-administered.
Self-reported quality of life | Baseline, once during with-robot phase, Week 5
  Participants will complete the RAND 36-Item Short Form Survey, which will be used to assess eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. All items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. Items in the same scale are averaged together to create the 8 scale scores. Scale scores represent the average for all items in the scale that the respondent answered.
Participant engagement with the robot | 2 weeks
  Visual analog scales, measured by the robot, will be analyzed to evaluate participant engagement during each of the ten 15-minute robotic assistance sessions that will occur over the course of two weeks.
Robot adherence | 2 weeks
  Robot adherence will be measured based upon attendance to the robotic assistance sessions. Each participant will be scheduled to attend ten robotic assistance sessions.
Dietary intake | Two 24-hour periods
  Dietary intake will be determined by two 24-hour diet recalls. One 24-hour recall will occur during the with-robot phase and the other will occur during the without-robot phase.
Program adherence | 5 weeks
  Adherence to the iDiet will be measured by the number videoconference sessions attended by the participant. Each participant will be scheduled to participate in six videoconference sessions (one/week), each one hour long.

CONTACTS AND LOCATIONS:
Overall Officials: Susan B Roberts, PhD, Principal Investigator — Tufts University Jean Mayer USDA Human Nutrition Research Center on Aging
Locations (1):
- Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salinardi TC, Batra P, Roberts SB, Urban LE, Robinson LM, Pittas AG, Lichtenstein AH, Deckersbach T, Saltzman E, Das SK. Lifestyle intervention reduces body weight and improves cardiometabolic risk factors in worksites. Am J Clin Nutr. 2013 Apr;97(4):667-76. doi: 10.3945/ajcn.112.046995. Epub 2013 Feb 20. PMID 23426035
- [Background] Briggs P, Scheutz M, Tickle-Degnen L, editors. Are Robots Ready for Administering Health Status Surveys': First Results from an HRI Study with Subjects with Parkinson's Disease. Proceedings of the Tenth Annual ACM/IEEE International Conference on Human-Robot Interaction; 2015: ACM.